CLINICAL TRIAL: NCT06929533
Title: Pharmacogenomics-Supported Psychotropic Prescribing Trial (PGx-SUPPORT): A Pilot Implementation Study in Manitoba
Brief Title: Pharmacogenomics-Supported Psychotropic Prescribing Trial
Acronym: PGx-SUPPORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: University of Calgary (Other); Shared Health Manitoba (Unknown); Winnipeg Regional Health Authority (Other); Health Sciences Centre, Winnipeg, Manitoba (Other)
Responsible Party: Principal Investigator, Abdullah Al Maruf, Assistant Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HS26637 (HS2024:279)
Record Dates: First submitted 2025-03-27; First posted 2025-04-16 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Mental Disorder; Pharmacogenetics; Adverse Drug Reaction (ADR); Effectiveness
Keywords: Adult; Mental Health; Psychiatry; Pharmacogenetics; Depression; Anxiety; OCD; Psychosis; Bipolar Disorder; mental illness
MeSH Terms: conditions — Mental Disorders; Drug-Related Side Effects and Adverse Reactions; Psychological Well-Being; Depression; Anxiety Disorders; Psychotic Disorders; Bipolar Disorder | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacogenetic Testing (Experimental): Pharmacogenetic testing panel (CYP2C19, CYP2D6, CYP2B6, CYP3A4, CYP3A5, CYP2C9, CYP4F2, DPYD, HLA-A, HLA-B, NUDT15, SLCO1B1, TPMT, VKORC1, 2C Cluster, UGT1A1)
  Interventions: Diagnostic Test: Pharmacogenetic Testing

INTERVENTIONS:
Diagnostic Test: Pharmacogenetic Testing — Participants will donate a 1ml (one-fifth of a teaspoon) sample of saliva. DNA extracted from the saliva sample will be used for genotyping. Genotyping results will be translated into an interpretative clinical report using evidence-based software (Sequence2Script) and delivered to the treating physician for use in their clinical decision-making. The report will contain genotyping results, predicted phenotype, and evidence-based drug selection and dosing recommendations relevant to the patient's current and future care.

SUMMARY:
Investigate the feasibility and utility of implementing pharmacogenetic testing for adults (aged 18 and older) seeking care for mental illness in Manitoba.

DETAILED DESCRIPTION:
Background and Rationale: Pharmacogenomic (PGx) testing utilizes genetic information as a surrogate marker of a person's ability to process and react to drugs. This information can be used to inform medication selection and dosing, reducing the number of trials needed to choose a suitable medicine. For Manitoba healthcare providers, the only access to psychiatric PGx testing is through commercial providers, costing patients $200 to $2,300. To the best of our knowledge, no study in Manitoba has previously evaluated the feasibility of PGx testing in adult patients seeking care for mental illness.

RESEARCH OBJECTIVES: We aim to investigate the feasibility and utility of implementing PGx testing in Manitoba for adult patients seeking care for mental illness.

Primary Outcome and Measures: Feasibility will be measured along four dimensions:

* Acceptability (satisfaction surveys - patient & clinician)
* Practicality (testing turnaround time)
* Implementation (clinicians' self-reported use of testing results in the prescribing decision-making process)
* Demand (number of referrals, clinicians' self-reported intent to use testing in the future)

Secondary Outcomes and Measures:

* Changes in global functioning and symptom severity [Clinical Global Impression (CGI) - Severity and Improvement; Brief Psychiatric Rating Scale (BPRS); DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure; Patient Health Questionnaire-9 (PHQ-9); General Anxiety Disorder-7 (GAD-7); Altman Self-Rating Mania Scale (ASRM); Early Psychosis Screener (EPS-26)]
* Adverse drug experience [Frequency, Intensity, Burden of Side Effects Rating (FIBSER)]
* Impact of PGx testing [Changes in medication prescribing and dispensing patterns; changes in healthcare utilization (e.g., inpatient length of stay, mental health resource use, and utilization of healthcare services)

Expected Outcomes: The findings from the proposed study will inform policymakers and facilitate decision-making and priority-setting related to implementing PGx-based psychotropic prescribing policies in Manitoba

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* The initiation, change, dose adjustment, or augmentation of psychotropic medication(s) is indicated
* The treating clinician thinks PGx testing can benefit and refers the patient to the study

Exclusion Criteria:

* Unwillingness to donate saliva samples for genetic analysis
* History of liver or bone marrow (hematopoietic cell) transplantation
* PGx testing results are already available
* No personal health identification number (PHIN) is available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Testing Acceptibility | 3 months after after baseline.
  Acceptability will be measured via a four-item patient satisfaction survey three months after the testing and a two-item clinician satisfaction survey after discharge. Responses will be recorded on a five-point Likert scale (1 = very dissatisfied to 5 = very satisfied).
Implementation Practicality | Up to 3 Months
  Practicality will be measured by the mean and median testing turnaround time (i.e., test ordering to return of results).
Implementation Feasibility | Patient discharge date [within 3 months of baseline].
  Implementation will be measured using a two-item clinician self-report questionnaire that asks about using testing results in the prescribing decision-making process. These will be Yes/No questions, with more "yes" responses indicating higher usefulness and interest in using the test in clinical practice.
Test Demands | Patient discharge date [within 3 months of baseline].
  Demand will be measured by the total number of referrals to the study and by a one-item clinician self-report questionnaire asking about intent to use the testing in the future. Responses will be recorded on a five-point Likert scale (1 = very unlikely to 5 = very likely).

SECONDARY OUTCOMES:
Clinical Global Impression Scale (CGI) - Severity | Baseline
  1 = normal, 7 = among the most extremely ill
Clinical Global Impression Scale (CGI) - Improvement | 3 months after baseline.
  Assesses the overall change in the patient's condition compared to baseline, on a 7-point scale (1 = very much improved, 7 = very much worse).
Brief Psychiatric Rating Scale (BPRS) | Baseline and patient discharge date, within 3 months.
  The rater enters a number for each symptom construct, ranging from 1 (not present) to 7 (extremely severe).
DSM-5-TR Self-Rated Level 1 Cross-Cutting Symptom Measure - Adult | Baseline and 3 months after baseline.
  This adult version of the measure consists of 23 questions that assess 13 psychiatric domains, including depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use. Each item on the measure is rated on a 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3=moderate or more than half the days; and 4=severe or nearly every day).
General Anxiety Disorder-7 (GAD-7) | Baseline and 3 months after baseline.
  This is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." GAD-7 total score for the seven items ranges from 0 to 21.
  0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Patient Health Questionnaire-9 (PHQ-9) | Baseline and 3 months after baseline.
  The PHQ-9 asks patients about the frequency with which they have experienced certain symptoms over the past two weeks, using a four-point scale (0 = "not at all" to 3 = "nearly every day"). The total score, ranging from 0 to 27, indicates the severity of depression, with higher scores suggesting more severe symptoms.
  Scoring:
  0-4: Minimal or no symptoms 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20 or higher: Severe depression
Altman Self-Rating Mania Scale (ASRM) - Adult | Baseline and 3 months after baseline.
  Each item on the measure is rated on a 5-point scale (i.e., 1 to 5) with the response categories having different anchors depending on the item. The ASRM score range from 5 to 25 with higher scores indicating greater severity of manic symptoms.
The Early Psychosis Screener (EPS-26) | Baseline and 3 months after baseline.
  The EPS-26 consists of 26 questions that assess for symptoms and experiences associated with psychosis. A higher score on the EPS-26 suggests a greater likelihood of being at risk for psychosis.
Frequency, Intensity, Burden of Side Effects Rating (FIBSER) | Baseline (if applicable) and 3 months after baseline.
  It measures three dimensions: the frequency of side effects, the intensity of these side effects, and the burden they impose on daily functioning. Each dimension is rated on a Likert scale, ranging from 0 to 6, where higher scores indicate greater severity and difficulty caused by side effects.
Healthcare Utlization | 1 year
  Changes in healthcare utilization (including inpatient length of stay) will be measured using a ten-item patient self-report mental health resource use questionnaire, medical charts, and administrative data records six months before and after the participant enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Al Maruf, PhD, M.Pharm., B.Pharm, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Shared Health Facilities, Winnipeg, Manitoba
  - University of Manitoba College of Pharmacy, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No